CLINICAL TRIAL: NCT03315260
Title: Treatment Satisfaction With Ra-223 Among Japanese Castration Resistant Prostate Cancer (CRPC) Patients
Brief Title: Treatment Satisfaction With Ra-223 in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19502
Record Dates: First submitted 2017-10-04; First posted 2017-10-20 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Prostatic Neoplasms
Keywords: Castration resistant prostate cancer; Patient reported outcome
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone metastatic CRPC patients: Japanese patients who are designated to undertake Ra-223/Xofigo therapy based on physician judgement
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Ra-223 is a radiopharmaceutical with an indication to treat Castration Resistant Prostate Cancer (approved indication in Japan)

SUMMARY:
This study aims to answer the research question: Are Japanese bone metastatic CRPC patients satisfied with their Ra-223 treatment, and what factors drive such satisfaction? It also aims to determine patient anxiety regarding prostate cancer while on treatment with Ra-223, and assess the effect on quality of life.

DETAILED DESCRIPTION:
This is a local, Japanese, prospective, longitudinal, observational, company-sponsored, multi-center, single arm study that will describe treatment satisfaction with Ra-223 in 150 bone metastatic CRPC patients on 1st to 3rd line CRPC therapy. All outcomes will be obtained using PRO questionnaires at 4 time points: before treatment, during treatment, and at 1-month after the last treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old (age of maturity in Japan)
* Male, diagnosed with CRPC
* With ≥2 bone metastases and no visceral metastasis based on the most recent imaging procedure
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) 0-1, not in end-stage palliative care
* Designated by examining physician to undergo Ra-223 treatment either in the 1st, 2nd, or 3rd line of CRPC therapy
* Has provided written, informed consent (in Japanese)
* Has ≥6 months life expectancy

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Currently receiving any chemotherapy for CRPC or any new hormone therapy (enzalutamide, abiraterone acetate) at enrolment
* Where any of the below conditions apply:

  * Started or switched to new androgen deprivation therapy (ADT) (e.g., LHRH agonists and antagonists, anti-androgens, estrogens,) within 4 weeks prior to enrolment or planning to start new treatment prior to 1st Ra-223 injection
  * Treatment with anticancer-chemotherapy within previous 4 weeks, or planned before the 1st Ra-223 injection, or failure to recover from adverse events (AEs) (CTCAE Grade >2) due to anticancer chemotherapy administered more than 4 weeks prior
  * Systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within the previous 24 weeks
  * Previous hemi-body external radiotherapy
* Imminent or established spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI)
* Presence of other maligancy at enrolment
* Otherwise deemed incapable of participating by examining physician

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese CRPC patients designated to receive Ra-223 (Xofigo)
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction with treatment using the Cancer Therapy Satisfaction Questionnaire (CTSQ) | From baseline to 7 months
  The CTSQ is a 16-item self-administered questionnaire measuring 3 domains related to patients' satisfaction with cancer therapy.

SECONDARY OUTCOMES:
Change in the total scores of the CTSQ domains | From baseline to 7 months
Change in patient anxiety with prostate cancer using the Memorial Anxiety Scale for Prostate Cancer (MAX-PC) | From baseline to 7 months
  Changes in the MAX-PC scores will be analyzed as full scores (no sub-domains).
Change in bone-related symptoms using the Functional Assessment of Cancer Therapy Quality of Life Measurement in Patients with Bone Pain (FACT-BP) | From baseline to 7 months
  Change in FACT-BP scores will be analyzed as full scores (no subdomains).
Differences in change in treatment satisfaction (measured by CTSQ) between potential subgroups | From baseline to 7 months
  Potential subgroups will be identified depending on the number of patients available for subgrouping.
Differences in change in prostate cancer anxiety (measured by MAX-PC) between potential subgroups | From baseline to 7 months
  Potential subgroups will be identified depending on the number of patients available for subgrouping.
Differences in change in bone pain (measured by FACT-BP) between potential subgroups | From baseline to 7 months
  Potential subgroups will be identified depending on the number of patients available for subgrouping.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Background] Akakura K, Uemura H, Kawakami S, Yokomizo A, Nakamura M, Nishimura K, Komori T, Ledesma DA. Metastatic castration resistant prostate cancer patients' experience with Radium-223 treatment in Japan. Future Oncol. 2024 Apr;20(12):781-798. doi: 10.2217/fon-2023-0870. Epub 2024 Jan 26. PMID 38275149